CLINICAL TRIAL: NCT01567462
Title: PK Button Vaporization Electrode for Treatment of Bladder Tumors
Brief Title: PlasmaKinetic (PK) Button Vaporization Electrode for Treatment of Bladder Tumors
Acronym: PK Button
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Kenneth Ogan, MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00053735; PK Button and Bladder Tumors (Other: Other)
Record Dates: First submitted 2012-03-27; First posted 2012-03-30 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-10

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; transurethral resection of bladder tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monopolar Electrocautery (Active Comparator): The current treatment standard of care for patients who present de novo or with a recurrent bladder tumor is transurethral resection of the bladder tumor (TURBT) using monopolar electrocautery in the form a 90-degree loop electrode and has been used since its introduction in 1952. This intervention, accomplished endoscopically through the urethra, is both diagnostic and potentially therapeutic. An adequately performed TURBT will provide the pathologist with enough tissue to provide tumor grade and stage information.
  Interventions: Device: Monopolar electrocautery loop in Transurethral resection of bladder tumors
- PK Button Vaporization Electrode (Active Comparator): Bipolar energy has been available for many years and has been readily adopted for the surgical treatment of benign prostatic enlargement and may provide advantages and solutions to the technical challenges of monopolar electrocautery. A further refinement on bipolar energy has been the recent introduction of the PlasmaKinetic (PK) Button Vaporization electrode which will be used in the intervention arm of this study. This electrode is already approved by the Food and Drug Administration (FDA) for this indication as well. The semi-spherical design of the electrode creates a plasma arc that glides over the tissue, transmitting energy to the cell layers adjacent to the arc which are then quickly vaporized.
  Interventions: Device: PK Button Vaporization Electrode in transurethral resection of bladder tumors

INTERVENTIONS:
Device: Monopolar electrocautery loop in Transurethral resection of bladder tumors — Standard monopolar electrocautery loop in transurethral resection of bladder tumors (TURBT)
  Arms: Monopolar Electrocautery
Device: PK Button Vaporization Electrode in transurethral resection of bladder tumors — PlasmaKinetic (PK) Button Vaporization Electrode in transurethral resection of bladder tumors (TURBT)
  Arms: PK Button Vaporization Electrode

SUMMARY:
The purpose of this study is to compare the use of two types of equipment during transurethral resection of bladder tumors (TURBT). The two types of surgical devices are: the monopolar loop electrocautery and the PlasmaKinetic (PK) Button Vaporization Electrode. These two devices do the same task but differ in the way they create electric current when removing cancerous tissue. The investigators hope to examine and compare the uses of these two surgical devices to see if any advantages do exist or whether they actually are similar. The goal of the study is to prove similarity in outcomes between the two techniques and analyze the outcomes resulting from each case.

DETAILED DESCRIPTION:
This study will study the medical intervention used when bladder cancer patients present with a new or recurrent bladder tumor. Currently when patients report these tumors, they undergo a standard practice called transurethral resection of the bladder tumor (TURBT) in order to determine the stage of the cancer. This intervention, accomplished by looking through the urethra using an endoscope, is both diagnostic and potentially therapeutic. An adequately performed TURBT will provide the pathologist with enough tissue to provide tumor grade and stage information. Currently, TURBT is done using equipment called monopolar electrocautery which is in the form a 90-degree loop electrode. Although usually safe and sufficient, this technique can create technical challenges because it can be difficult to position the loop electrode in a dynamically changing cylindrical space (the bladder). Specifically, especially with larger bladder tumors, intraoperative bleeding can obscure visualization and result in incomplete tumor resection as well as inadequate sampling of the layers of the bladder needed to establish tumor stage. Furthermore, monopolar current can result in stimulation of a nerve (the obturator nerve) during resection of wall tumors, resulting in violent movement of the leg which can cause a potential bladder tear as well as possible (iliac) vessel injury.

Conversely, a technique using bipolar energy, which has been available for many years, has been readily adopted for the surgical treatment of benign prostatic enlargement. The advantages of a bipolar electrical current include the direct return of electrical current to the loop rather than to a grounding pad placed on the patient's skin. This has the theoretical value of limiting the diffusion of electrical current, and therefore heat, to the surrounding tissue. A further refinement on bipolar energy has been the recent introduction of a piece of equipment called the PlasmaKinetic (PK) Button Vaporization electrode, which is currently approved by the Food and Drug Administration (FDA) for this indication. Coupling bipolar energy into the Button electrode would not only harness the benefits of less thermal spread but also would obviate the geometric challenges associated with loop electrodes during resection of bladder tumors. Procedural advantages would potentially include minimal bleeding, good visualization, and a reduction in the occurrence of the obturator reflex and concomitant bladder perforation.

This study is a randomized double-arm trial examining the results of both techniques for bladder cancer TURBT procedures with a minimum of 120 patients at Emory. The purpose of this study is to measure the procedural (intraoperative), short term, as clinically indicated (4-6 weeks), and long-term (3 months) outcomes of TURBT using the PK Button when compared to traditional monopolar loop electrocautery. The goal of the study is to prove equivalence in outcomes between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystoscopically detected bladder tumors requiring TURBT
* Patients with bladder tumors which are endoscopically resectable by surgeon's judgment with only one trip into the operating room.

Exclusion Criteria:

* Patients with clinical evidence of locally advanced, nodal, or metastatic bladder cancer
* Patients with hydronephrosis secondary to bladder cancer
* Patients with diffuse tumor throughout bladder that is deemed unresectable by surgeon

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ogan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Urology, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between September 2012 and March 2017. Of the 95 participants who signed consent, 90 subjects began study participation.
Groups:
- Monopolar Loop Electrocautery: Participants underwent a transurethral resection of the bladder tumor (TURBT) using monopolar loop electrocautery.
- PK Button Vaporization Electrode: Participants underwent a transurethral resection of a bladder tumor using a PK button vaporization electrode.
Period: Overall Study
Arm/Group | Monopolar Loop Electrocautery | PK Button Vaporization Electrode
Started | 45 | 45
Completed | 41 | 38
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 4 | 7

BASELINE CHARACTERISTICS:
Population: Participants who completed all study procedures per protocol.
Groups:
- Monopolar Loop Electrocautery: Participants completed a transurethral resection of the bladder tumor (TURBT) using monopolar loop electrocautery and all follow up procedures.
- PK Button Vaporization Electrode: Participants completed a transurethral resection of a bladder tumor using a PK button vaporization electrode and all follow up procedures.
- Total: Total of all reporting groups
Arm/Group | Monopolar Loop Electrocautery | PK Button Vaporization Electrode | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (12.2) | 69.2 (11.4) | 69 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 29 | 30 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 22 | 46
  Non-White | 7 | 7 | 14
  Unreported | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 38 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Procedural Complications
Description: The number of procedural complications describes the total number of post-operative bleeding, need for blood transfusion, bladder perforation, obturator nerve stimulation, catheterization time, or need for hospitalization or bladder irrigation events that occur within thirty days of the procedure.
Time Frame: Post-Intervention (Up to 30 Days)
Population: Participants who completed all study procedures per protocol.
Measure: Number; unit: complications
Arm/Group | Monopolar Loop Electrocautery | PK Button Vaporization Electrode
Number analyzed (Participants) | 41 | 38
complications | 23 | 15

2. Secondary Outcome: Mean Operative Time
Description: The average operative time was measured through study completion.
Time Frame: After Surgery Completion, Up to 174 Minutes
Population: Participants who completed all study procedures per protocol.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Monopolar Loop Electrocautery | PK Button Vaporization Electrode
Number analyzed (Participants) | 41 | 38
minutes | 46.0 (28.7) | 56.4 (35.4)

3. Secondary Outcome: Mean Catheterization Time
Description: The average duration of the catheterization time was measured through study completion.
Time Frame: After Surgery Completion, Up to 336 Hours
Population: Participants who required catheterization after the operative procedure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Monopolar Loop Electrocautery | PK Button Vaporization Electrode
Number analyzed (Participants) | 40 | 35
hours | 46.7 (74.9) | 45.9 (72.9)

4. Secondary Outcome: Number of Participants With Disease Recurrence
Description: The number of participants who had disease recurrence within the four month follow up period.
Time Frame: Post-Intervention (Up to 4 Months)
Population: Participants who completed all study procedures per protocol.
Measure: Number; unit: participants
Arm/Group | Monopolar Loop Electrocautery | PK Button Vaporization Electrode
Number analyzed (Participants) | 41 | 38
participants | 8 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (5 years).
Arm/Group | Monopolar Loop Electrocautery | PK Button Vaporization Electrode
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 5/45 | 1/45
Other Adverse Events (participants affected / at risk) | 11/45 | 4/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monopolar Loop Electrocautery (N=45) | PK Button Vaporization Electrode (N=45)
Postoperative Bleeding (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Bladder Perforation (Renal and urinary disorders) | 5 (5) | 0 (0)
Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monopolar Loop Electrocautery (N=45) | PK Button Vaporization Electrode (N=45)
Continuous Bladder Irrigation (Injury, poisoning and procedural complications) | 11 (11) | 4 (4) — Need for continuous bladder irrigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT01567462/Prot_SAP_000.pdf